CLINICAL TRIAL: NCT07017335
Title: A Phase 1 Clinical Trial to Evaluate the Drug-Drug Interaction Between R1_PBK_M2301 and R2_PBK_M2301
Brief Title: Drug-Drug Interaction Between R1_PBK_M2301 and R2_PBK_M2301 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PBK_M2301_101
Record Dates: First submitted 2025-05-23; First posted 2025-06-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Drug-Drug Interaction Healthy Volunteers
Keywords: Drug-Drug Interaction; Levodropropizine; Pelargonium sidoides; Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group, open-label, Phase 1 study to evaluate the drug-drug interaction (DDI) between R1_PBK_M2301 (levodropropizine) and R2_PBK_M2301 (Pelargonium sidoides dry extract) in healthy adult volunteers. Participants will be assigned to two arms to receive either R1_PBK_M2301 or R2_PBK_M2301 followed by co-administration, in parallel design.
Masking Description: This is an open-label study. No parties, including participants, investigators, or outcomes assessors, are masked to intervention assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R1_PBK_M2301 Administration (Experimental): Participants in this arm will receive R1_PBK_M2301, which contains 60 mg of levodropropizine per tablet, to evaluate drug-drug interactions.
  Interventions: Drug: R1_PBK_M2301(Levocloperastine 60mg)
- R2_PBK_M2301 Administration (Experimental): Participants in this arm will receive R2_PBK_M2301, which contains 20 mg of Pelargonium sidoides ethanol extract (11%) per tablet, to evaluate drug-drug interactions.
  Interventions: Drug: R2_PBK_M2301 (Pelargonium sidoides extract)

INTERVENTIONS:
Drug: R1_PBK_M2301(Levocloperastine 60mg) — R1_PBK_M2301 is a test drug containing 60mg of levocloperastine per tablet. It is administered orally to evaluate pharmacokinetic characteristics and potential drug-drug interactions with R2_PBK_M2301 in healthy adult volunteers.
  Arms: R1_PBK_M2301 Administration
Drug: R2_PBK_M2301 (Pelargonium sidoides extract) — R2_PBK_M2301 is an oral tablet containing 20 mg of Pelargonium sidoides 11% ethanol extract, used as a comparator to evaluate potential pharmacokinetic interactions with R1_PBK_M2301.
  Arms: R2_PBK_M2301 Administration

SUMMARY:
This is a Phase 1, open-label, randomized, crossover clinical trial designed to evaluate the potential drug-drug interaction (DDI) between R1_PBK_M2301 (levodropropizine 60 mg) and R2_PBK_M2301 (Pelargonium sidoides ethanol extract 11%) in healthy adult volunteers. The study aims to assess the pharmacokinetics of each investigational drug when administered alone and in combination. Approximately [insert number] healthy subjects will participate in two treatment periods with appropriate washout intervals. Safety, tolerability, and pharmacokinetic parameters will be evaluated to support future combination development.

DETAILED DESCRIPTION:
This Phase 1 clinical trial is designed to assess potential drug-drug interactions between R1_PBK_M2301 (levodropropizine 60 mg) and R2_PBK_M2301 (Pelargonium sidoides 11% ethanol extract) in healthy adult volunteers. The study adopts an open-label, randomized, two-period crossover design. Each participant will receive both investigational products in different periods, with a washout interval between treatments.

The primary objective is to compare the pharmacokinetic parameters (e.g., C_max, AUC) of the individual drugs when administered alone versus in combination. Secondary objectives include evaluating safety and tolerability through clinical assessments, vital signs, ECGs, and laboratory tests.

Approximately 24 healthy adults will be enrolled. Each subject will be screened for eligibility based on predefined inclusion and exclusion criteria. Eligible participants will be randomly assigned to one of two sequence groups. Blood samples will be collected at predetermined time points to analyze plasma concentrations of the study drugs.

The findings of this study are expected to support further clinical development and regulatory planning for the combination use of levodropropizine and Pelargonium sidoides extract.

ELIGIBILITY:
<Inclusion Criteria>

1. Healthy male or female adults aged ≥19 and <65 years at the time of screening.
2. Body mass index (BMI) between 18 and 30 kg/m² (BMI = weight [kg] / height² [m²]);

   * Male participants must weigh at least 50 kg.
   * Female participants must weigh at least 45 kg.
3. No clinically significant congenital or chronic diseases, and no abnormal findings from a medical examination (e.g., electroencephalogram, electrocardiogram, chest and/or gastrointestinal endoscopy, or radiologic examinations, if deemed necessary).
4. Laboratory test results (including hematology, clinical chemistry, coagulation tests, serology, urinalysis) and ECG results deemed suitable for study participation by the investigator (or sub-investigator).
5. Willing and able to voluntarily provide written informed consent after receiving detailed information about the study, and agrees to comply with study requirements.
6. Agrees to use medically accepted contraception methods* from the first administration of the investigational product through 1 week after the final administration, and agrees not to donate sperm or ova during this period.

   * Medically accepted contraception includes intrauterine devices (IUD, IUS), sterilization (vasectomy or tubal ligation), or combination of barrier methods (e.g., male/female condoms, cervical caps, diaphragms, sponges), possibly with spermicide.

<Exclusion criteria>

1. Use of enzyme-inducing or enzyme-inhibiting drugs such as barbiturates within 30 days prior to the first dose, or use of any medication that may interfere with the study within 10 days prior to the first dose.
2. Participation in another clinical trial involving administration of an investigational drug or bioequivalence study within 6 months prior to the first dose.
3. Donation of whole blood within 8 weeks, donation of blood components within 2 weeks, or receipt of blood transfusion within 4 weeks prior to the first dose.
4. History of gastrointestinal surgery that may affect drug absorption (excluding appendectomy and hernia repair).
5. Within 1 month prior to the first dose, meets one of the following:

   * Alcohol consumption >21 drinks/week (males) or >14 drinks/week (females);

     (1 drink = 50 mL soju, 250 mL beer, or 30 mL whiskey)
   * Smoking >20 cigarettes/day on average.
6. Individuals with any of the following conditions:

   * Known hypersensitivity to the investigational product or its components
   * Increased bronchial mucus secretion
   * Mucociliary dysfunction (e.g., Kartagener syndrome, primary ciliary dyskinesia)
   * Bleeding tendency or use of anticoagulants
   * Severe hepatic impairment
   * Severe liver or kidney disease
   * Genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
7. History of clinically significant psychiatric illness.
8. Any other condition deemed by the principal investigator (or sub-investigator) to render the subject unsuitable for study participation.
9. Female participants who are pregnant, suspected of being pregnant, or breastfeeding.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of R1_PBK_M2301 and R2_PBK_M2301 | Up to 48 hours post-dose per treatment period
  Evaluation of potential pharmacokinetic interaction between R1_PBK_M2301 and R2_PBK_M2301 by comparing Cmax values after single oral administration alone and in combination in healthy adult subjects.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC₀-t) | Up to 48 hours post-dose per treatment period
  Evaluation of potential pharmacokinetic interaction between R1_PBK_M2301 and R2_PBK_M2301 by comparing AUC₀-t values after single oral administration alone and in combination in healthy adult subjects.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC₀-∞) | Up to 48 hours post-dose per treatment period
  Evaluation of potential pharmacokinetic interaction between R1_PBK_M2301 and R2_PBK_M2301 by comparing AUC₀-∞ values after single oral administration alone and in combination in healthy adult subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- H+ Yangji Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to internal policy and data protection regulations. The dataset is limited to a small population of healthy volunteers and is intended solely for internal analysis and regulatory submission.